CLINICAL TRIAL: NCT04346992
Title: Prevalence Of Keratoconus Among Patients With Thyroid Gland Dysfunction
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Omar Said, Dr, Fayoum University
Other Study IDs: R109
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Keratoconus in Thyroid Gland Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: blood sample to measure thyroid profile
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Hormonal imbalances are likely to affect the corneal metabolism and may be also associated with Keratoconus. Among the various endocrinologic dysfunctions assumed so far, thyroid gland dysfunction (TGD) (hypo- or hyperthyroidism; comprised as TGD) is frequently associated with eye diseases such as Graves disease

DETAILED DESCRIPTION:
Aim of the work

We aim to examine the prevalence of KC among patients already diagnosed by endocrinologist with TGD.

Materials and methods

Our Screening for KC will include evaluation of the demographic data and complete ophthalmological examination of the patients using:

VA Refraction K reading Slit lamp examination Pentacam Study design Epidemiological study

Inclusion citeria All patients diagnosed as thyroid gland dysfunction Control group

Exclusion criteria Uncooperative patients

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as thyroid gland dysfunction

Exclusion Criteria:

* Uncooperative patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: we will enroll all patients who meet the inclusion criteria and signed a written informed consent form
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
prevalence of keratoconus in thyroid gland dysfunction | we will recruit patients who meer the inclusion criteria during the study period April-August 2020
  Our Screening for KC will include evaluation of the demographic data and complete ophthalmological examination of the patients using:
  VA Refraction K reading Slit lamp examination Pentacam

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No